CLINICAL TRIAL: NCT03210870
Title: Clatsop Astoria Maternal Partnership Study (CAMPS) - Healthy Eating in Pregnancy Intervention
Acronym: CAMPS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan Purnell, Professor and Associate Director, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00011099
Record Dates: First submitted 2017-05-25; First posted 2017-07-07 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Pregnancy Related
Keywords: Maternal health; maternal nutrition; fetal health related to maternal nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Other): In-person nutritional education classes
  Interventions: Behavioral: nutritional education classes
- Control (No Intervention): no in-person nutritional education classes

INTERVENTIONS:
Behavioral: nutritional education classes — The objective to be accomplished through the completion of a nutritional education program for pregnant women that incorporates the biopsychosocial principles of the Satter Eating Competence Model. Emphasizing healthy food choices and improve eating competency.
  Arms: Intervention

SUMMARY:
Purpose of this study is to learn more about how nutritional advice given during pregnancy affects a mother's food choices and her baby's growth.

DETAILED DESCRIPTION:
The overall goal of this proposal is to effect change in women's nutritional behaviors that will improve not only their own health and that of their unborn child. Because solutions and needs for prevention of chronic diseases are unique and especially challenging for rural areas, we have chosen to stage our studies in the northern coast of Oregon, centered on the town of Astoria.

Our objective is to assess the effect on markers of maternal health and fetal growth of providing education that includes the rationale and practical aspects of healthy cooking during pregnancy to improve her baby's lifetime risk for cardiovascular disease and other chronic diseases. We will accomplish this objective through the completion of a nutritional education program for pregnant women that incorporates the biopsychosocial principles of the Satter Eating Competence Model in the curriculum, including:

* Emphasizing healthy food choices:

  1. Whole foods
  2. Plant-based (fruits, vegetables, plant-based oils/fats) and whole grains
  3. Fish and lean meats
  4. Non-fat dairy
* Avoiding / minimizing intake of unhealthy foods, such as processed foods/meals and sugar-added beverages
* Improving eating competency by:

  1. Developing and maintaining positive attitudes about eating and food
  2. Acceptance skills that support eating an ever-increasing variety of the available food
  3. Following internal regulation signals that allow intuitively consuming enough food to give energy and stamina and to support stable body weight
  4. Enhancing skills and resources for orchestrating family meals

  3. Background

Developmental Origins of Health and Disease There is increasing evidence that the health of adult populations is influenced by the nutritional provision imparted to its members during their conception and through the first three years of their post-conception life, reflecting the origination of the structures in an individual's body from developmental processes. The links between early nutrition and later health initially came to light through the work of Dr. David Barker, who showed that in poorer regions of the UK, those who survived infancy predominantly died of athersclerotic disease as adults and demonstrated an inverse relationship between birthweight and ischemic heart disease. Similar relationships between low birth weights with increased risk of heart disease have now been replicated in the United States, Scandinavian countries, Finland, the Netherlands and in India, as well as in animal models of nutritional deprivation.

Subsequent research has demonstrated that people who grew poorly before birth or as infants are at risk not only for heart disease but also for other adult chronic diseases including hypertension, type 2 diabetes, obesity, asthma, and osteoporosis. Poor growth in early life has also been associated with compromised cognitive function. It is now believed, based on animal and human data that prenatal stressors in the form of nutrition, high levels of stress hormone (cortisol), and hypoxia lead to structural and epigenetic changes that impart vulnerability for disease in later life. The developmental response to these stressors is known as "programming," or the developmental origins of adult diseases.

While the original work in this field focused on maternal undernutrition as a source of stress for the developing baby, animal and human data suggest that exposure to a maternal diet that is calorically "sufficient" but of low-quality foods, such as the consumption of increasingly processed foods by Western societies, can result in similar in-utero programing and predisposition to obesity, diabetes, and cardiovascular disease in offspring. Especially concerning about these findings is the implication that reversal of these effects will take generations to realize. "Transgenerational nutritional flow" occurs because the eggs that will be fertilized to form babies in women of child-bearing age today began development in the ovaries of their mothers when their mothers were themselves in their grandmothers' womb. Thus the grandmother not only provided for the health of her own eggs, which became the mother, but also supplied the nutrients for the reproductive organs (including ovaries) in the mother as she developed from fetus to baby, thereby influencing the programming of her future grandchildren. Thus, we can now link the health status of the current citizens of Oregon with generational nutritional flow over the past century. Fortunately, evidence shows that improving the environment of mothers-to-be by lowering stress and providing access to healthier foods can reverse many of the adverse effects that are programmed in early life, though the full benefits of these efforts will take generations to realize.

The serious nature of these findings is evident by virtually any indicator of current population health in America, which point to a dramatic worsening over the last two decades with increasing rates of obesity and type 2 diabetes among adults and children, greater numbers of people with uncontrolled hypertension, increasing hospitalization rate of for heart failure, and ever decreasing birthweight. Recent studies predict further increases in these chronic disease rates based on current indicators. Such disease rates will make health care financially unsustainable. Worsening diets of mothers in recent decades has most certainly contributed to the deteriorating health status of Oregonians, mandating that novel innovations in dietary interventions are needed to bring wholesome nutrition to large segments of the population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Early pregnancy (6-14 weeks)
* Fluent in English

Exclusion Criteria:

* Failure to provide informed consent
* Active smokers or recreational drug users (including excessive alcohol defined as > 2 drinks per day)
* Circumstances that would prevent participation in group classes and study-related activities
* Diagnosis of type 1 or gestational diabetes at the time of entry
* Moving away from the local area in less than 1 year
* Planned delivery at a hospital other than Columbia Memorial Hospital in Astoria, Oregon

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in Heathy Eating Index Score (HEI) | The duration of study participation will last from early pregnancy through 6 months after delivery
  The primary outcome will be the change in healthy eating index (HEI) score obtained from the food frequency questionnaire as a result of assignment to the nutrition intervention or usual care. This outcome will be assessed at three time points: at baseline (~ 8 to 10 weeks gestation), after completion of the intervention (~ 20 to 24 weeks), and 6-months postpartum.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Q Purnell, MD, Principal Investigator — OHSU Knight Cardiovascular Institute
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No